CLINICAL TRIAL: NCT01096173
Title: Determination of the in Vitro Effects of CALM on COPD Sputum
Brief Title: Determination of the in Vitro Effects of Cationic Airway Lining Modulators (CALM) on Chronic Obstructive Pulmonary Disease (COPD) Sputum
Status: Completed | Type: Observational
Sponsor: Pulmatrix Inc. (Industry)
Collaborators: The VA Western New York Healthcare System (U.S. Federal Agency); Buffalo Institute For Medical Research (Unknown)
Responsible Party: Dr. Sanjay Sethi, MD, VA of Western NY Healthcare System, Buffalo Institute for Medical Research
Other Study IDs: PUL_VABUF_01
Record Dates: First submitted 2010-03-25; First posted 2010-03-30 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Sputum; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Biospecimen Retention: None Retained — Sputum samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is intended to be an evaluation of the properties of human sputum collected from patients with COPD. It is hypothesized that cationic airway lining modulators will have beneficial effects on the rheological properties of sputum derived from patients with COPD. Approximately 10 patients with COPD will collect sputum at home for 5 days. Samples will be collected and tested in laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and spirometric diagnosis of COPD
2. Smoking history of at least 10 pack yrs
3. Sputum production of greater than 2 tablespoons per day by patient report.

Exclusion Criteria:

1. a primary diagnosis of asthma or bronchiectasis
2. a COPD exacerbation within 4 weeks
3. Inability to comply with study procedures.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic setting
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sethi, MD, Principal Investigator — Va Western NY Healthcare, Buffalo Institute for Medical Research
Locations (1):
- VA WNY Healthcare System, Buffalo, New York, United States